CLINICAL TRIAL: NCT02572583
Title: A Clinical Study of Treating Influenza With Liugan Shuangjie Heji
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013BAI13B021
Record Dates: First submitted 2015-04-12; First posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-04

CONDITIONS: Influenza
Keywords: Reconciling Exterior and Interior Therapy; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — shufeng jiedu; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liugan Shuangjie Heji Group (Experimental): Liugan Shuangjie Heji, take orally, 4 times a day, 100 ml each time (i.e. two doses per day), for a course of five days.
  Interventions: Drug: Liugan Shuangjie Heji
- Shufeng Jiedu Capsule Group (Active Comparator): Shufeng Jiedu Capsule, take orally, 3 times a day, 4 capsules each time, for a course of five days.
  Interventions: Drug: Shufeng Jiedu Capsule
- Oseltamivir Phosphate Capsule Group (Active Comparator): Oseltamivir Phosphate Capsule, take orally, 2 times a day, 75 mg each time, for a course of five days.
  Interventions: Drug: Oseltamivir Phosphate Capsule

INTERVENTIONS:
Drug: Liugan Shuangjie Heji
  Arms: Liugan Shuangjie Heji Group
Drug: Shufeng Jiedu Capsule
  Arms: Shufeng Jiedu Capsule Group
Drug: Oseltamivir Phosphate Capsule
  Arms: Oseltamivir Phosphate Capsule Group

SUMMARY:
This prospective randomized controlled trial studies the efficacy and safety of treating influenza with the reconciling exterior and interior therapy. A total of 300 cases of seasonal flu in Beijing is to be collected, and divided into one treatment group and two control groups. Patients in the treatment group will receive Liugan Shuangjie Heji, while patients in control groups will receive Shufeng Jiedu Capsule and Oseltamivir Phosphate Capsule respectively, for a course of 5 days. The study assesses the efficacy and safety of treating influenza with the reconciling therapy based on the following outcome measures: the time it takes from the medicine intake to 0.5℃ drop of body temperature, and the time it takes for the body temperature to return to normal.

ELIGIBILITY:
Inclusion Criteria:

1. The disease in flu season of flu, in line with the western medicine clinical diagnostic criteria for influenza;
2. All influenza patients with TCM syndrome differentiation for the table is cold in the exterior and heat in the interior;
3. The course of the disease within 48 hours, the axillary temperature is 38.0 degree or higher;
4. Aged between 18 to 65 years;
5. Voluntary and signed informed consent.

Exclusion Criteria:

1. The first time to see a doctor Have used traditional Chinese medicine, or antiviral drugs;
2. Routine blood WBC is greater than the upper limit of normal;
3. Chest X-ray examination with inflammatory exudation images;
4. With cardiovascular, liver, kidney and hematopoietic system such as severe primary disease, immunodeficiency disease, cancer, mental illness, without self-knowledge, liver and kidney function significantly abnormal liver meritorious service is more than 1.5 times higher than normal;
5. Pregnancy, nursing mothers, and allergic constitution;
6. Participated in clinical subjects for nearly three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
time from the medicine intake to 0.5℃ drop of body temperature | five days
time for the body temperature to return to normal | five days

CONTACTS AND LOCATIONS:
Overall Officials: Yang - Jiao, MD, Study Director — Dongfang Hospital Beijing University of Chinese Medicine
Locations (1):
- Dongfang Hospital affiliated to Beijing University of Chinese Medicine, Beijing, China